CLINICAL TRIAL: NCT04437446
Title: OCT Angiography in the Glaucoma Diagnosis : A Multicenter Study
Brief Title: OCT Angiography in the Glaucoma Diagnosis
Acronym: OCTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OCTA
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Glaucoma
Keywords: Glaucoma; OCT; OCTA
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: The study is a prospective multicentric and interventional trial that aims to compare the vascular density between patients with glaucoma and patients without glaucoma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case Group (Experimental): The "Case" group corresponds to patients with glaucoma following the clinical criteria for glaucoma:
  * papilla excavation> 5/10 with altered ISNT rule, or neuro-retinal rhyme characteristic of glaucoma, or fiber alterations characteristic of glaucoma.
  * OCT with typical alterations (loss of the layer of nerve fibers or loss of these ganglion cells), loss of fibers typical of glaucoma.
  * Humphrey 24: 2 visual fields produced, reliable and typical of glaucoma.
  The assignment to the "Cas" group will be carried out by an ophthalmologist specializing in glaucoma according to the following criteria:
  - The intraocular pressure must be increased before the start of treatment (21 mmHg or more), except in cases of normal pressure glaucoma.
  The additional examination corresponds to an OCTA alone leading to an extension of the duration of the consultation by 5 minutes.
  Interventions: Diagnostic Test: Case Group
- Control Groupe (Experimental): The Control group corresponds to patients with no glaucoma, no suspicion or history of glaucoma, ocular hypertension, or alterations detected during the ophthalmological consultation.
  Witnesses will be matched to cases by age (+/- 5 years) and gender.
  For patients in this group, the additional examinations correspond to a visual field, an OCT and an OCTA leading to an extension of the duration of the consultation by 35 minutes.
  Interventions: Diagnostic Test: Control Group

INTERVENTIONS:
Diagnostic Test: Case Group — The additional examination corresponds to an OCTA which is a non-invasive examination, without potential risks, without radiation, using infrared light.
  Arms: Case Group
Diagnostic Test: Control Group — The additional examinations correspond to:
  * OCTA which is a non-invasive examination, without potential risks, without radiation, using infrared light.
  * OCT: non-invasive examination, without potential risks, without radiation, using infrared light. The patient must sit in front of a screen and a contact is taken without contact in about ten seconds.
  * Visual field
  Arms: Control Groupe

SUMMARY:
Glaucoma is a chronic degenerative disease of the optic nerve. It is the second cause of blindness worldwide and a frequent cause of irreversible blindness. In 2020, epidemic health authorities have predicted about 80 million glaucoma patients. Glaucoma can be treated by topical treatment (eye drops), laser or surgery. A premature diagnosis of glaucoma is very important to prevent irreversible blindness. Pachymetry, Optical Coherence Tomography (OCT) and visual fields exams are fundamental for the development of the glaucoma diagnosis. The severity of glaucoma is defined with Hodapp-Parrish-Andersen visual field criteria. According to these criteria, glaucoma can be classified as early (with average visual field deviation, MD, of 0 to -6 dB), moderate (MD of -6 to -12 dB) and severe (MD worse than -12 dB). The progression of glaucoma is being identified by the visual fields tests, and also by the progression of alterations in the optic nerve head. The visual fields tests are long and difficult (30 minutes). It is therefore important to create additional tests and anticipate the diagnosis, in order to avoid the irreversibility of glaucoma.

DETAILED DESCRIPTION:
The OCT Angiography (OCTA) is a non-invasive technology, marketed since 2014, that uses OCT with infrared light, with no radiation nor side effects, to evaluate within seconds the vascularization of the fundus, retina and optic nerve head, which may be useful for the glaucoma diagnosis. A recent meta-analysis has shown a decrease of the vascular density (DV) in glaucoma, so that OCTA may be useful in the advanced diagnosis of glaucoma. However, the VD values obtained were different depending on the device. In addition, no studies with the OCT Triton (Topcon®) device were considered in the analysis. The authors suggested the development of dedicated software, which would allow the evaluation of VD with different devices for a more independent and valid assessment. On the other hand, recent studies show that the diagnostic capacity of OCTA may be superior to that of OCT, and that OCTA may be more useful in determining the severity of glaucoma than OCT. It is therefore necessary to evaluate the additional diagnostic tests whether they are non-invasive and whether it allow us to give a faster diagnosis.

This study is aimed at comparing the diagnostic utility of OCTA with standard complementary glaucoma examinations (OCT and CV).

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient consultant in the ophthalmology department of the Marie-Thérèse Health Center or the Polyclinique de la Baie
* French speaking patient
* Patient affiliated to a health insurance plan
* Patient having given free, informed and express consent

Exclusion Criteria:

* Patient with another ophthalmological pathology or a history of ophthalmological pathology
* Patient with a history of ophthalmic surgery except for uncomplicated cataract surgery
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Vascular density between the 2 groups | Day1
  This outcome corresponds to percentage of vascularization of the optic papilla measured using OCTA.

SECONDARY OUTCOMES:
Papilla supply according to severity of glaucoma | Day 1
  This outcome corresponds to the comparison of the percentages of vascular density as a function of the severity of glaucoma.
Difference of papilla vascularization depending on the regions of the papilla | Day 1
  This outcome corresponds to the comparison of the percentages of vascular density as a function of the regions of the papilla (intra-papillary, peripapillary, superior, inferior, nasal, temporal).
  184/5000 corresponds to the comparison of the percentages of vascular density as a function of the regions of the papilla (intra-papillary, peripapillary, superior, inferior, nasal, temporal).
Vascularization of different regions of the papilla between case patients and control patients | Day 1
  This outcome corresponds to the comparison of the percentages of vascular density of the regions of the papilla between the case patients and the control patients.
Evaluation of the diagnostic performance of OCTA | Day 1
  This outcome corresponds to the comparison of the sensitivity and the specificity of OCTA compared to the additional examinations conventionally carried out within the framework of the diagnosis of glaucoma (OCT and visual fields) within the various regions of the vascular papilla between the case patients and the control patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yves LACHKAR, MD, Study Director — Fondation Hôpital Saint-Joseph
Locations (2):
- France (2):
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - Polyclinique de la Baie, Saint-Martin-des-Champs